CLINICAL TRIAL: NCT01279759
Title: Pre- and Post Operative Predictive Factors for Function 6 Months After Anterior Cruciate Ligament Reconstruction
Brief Title: Follow up of Patients Operated With Anterior Cruciate Ligament Reconstruction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haraldsplass Deaconess Hospital (Other)
Collaborators: University of Bergen (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Other Study IDs: 01339
Record Dates: First submitted 2010-11-08; First posted 2011-01-19 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Anterior Cruciate Ligament Reconstruction Predictive Factors; Function Downstairs walking Step time Symmetry

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

An estimated 4000 Anterior Cruciate Ligament Injuries (ACL) occur annually in Norway (Granan et al., 2004). 1630 primary ACL reconstructions were performed in Norway in 2008 (Norwegian Arthroplasty Register, 2009). Approximately 120 of these ACL reconstructions were performed at Haraldsplass Deaconess Hospital.

Physical therapists at our hospital are responsible for postoperative outpatient controls of patients with a reconstructed anterior cruciate ligament. A clinical observation is that stair walking (especially downstairs) may be problematic up to 6 months after ACL reconstruction. One reason may be that the quadriceps muscle is unable to control the knee when the subject is walking downstairs, and that the knee is perceived to be unstable. Other contributing factors may be pain and swelling.

It is of interest to know which pre and post operative factors can predict measured and patient reported function 6 months after ACL reconstruction. Previous research shows that predictive factors for clinical outcome after ACL reconstruction are anterior knee pain (Heijne et al., 2009), preoperative electromyography, early postoperative strength (McHugh et al., 2002), preoperative quadriceps muscle strength deficits, meniscus injury and pain (Eitzen et al., 2009), obesity, smoking and serious chondrosis (Kowalchuk et al., 2009).

Purpose:

1. To analyse which pre and post operative factors can predict measured and patient reported function 6 months after Anterior Cruciate Ligament reconstruction.
2. To investigate if there is an asymmetry in step time between the affected and unaffected leg during down stairs walking, and if degree of asymmetry decreases during a 6 months period post operatively. Further we want to compare step time asymmetry with other established outcome measures to investigate sensitivity to change over the observation period and also compare the patient group in this study with a control group of healthy subjects to see if asymmetry in the patient group after 6 months is still higher than in healthy subjects.

DETAILED DESCRIPTION:
Methods:

The investigators wish to recruit 35 people scheduled for anterior cruciate ligament (ACL) reconstruction with hamstrings tendon graft.

Patients will be asked to write a training diary.

Data will be collected 1 day preoperatively, 2 days, 6 weeks, 3 months and 6 months post operatively.

Ethics:

All participants will have to give informed consent before inclusion. All information obtained through the surveys will be treated confidentially. Participation is completely voluntary.

References:

GRANAN, L., ENGEBRETSEN, L. & BAHR, R. (2004) Kirurgi ved fremre korsbåndskader i Norge - sett fra et idrettsmedisinsk perspektiv. Tidsskr Nor Lægeforen, 124, 928-930.

NASJONALT REGISTER FOR LEDDPROTESER (2009) Nasjonalt korsbåndregister. Ortopedisk klinikk Haukeland Universitets Sykehus.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for reconstruction of the anterior cruciate ligament with hamstrings graft at Haraldsplass Deaconess hospital.

Exclusion Criteria:

* Patients with multiligament tears, meniscus suture, other problems that can influence strength testing, functional testing and gait symmetry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients planned for reconstruction of the anterioir crucuate ligament with hamstrings graft.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2010-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Asymmetry in step time between the affected and unaffected leg during down stairs walking. | 6 months postoperatively
  A triaxial kinematic sensor (XSens Mtx) positioned at the level of the lower trunk will be used to identify foot strike and separate left and right steps.
Isokinetic muscle strength measured with a fixed dynamometer (isok BI con/con 60/60 240/240 BIODEX). | 6 months postoperatively
Single leg hop test for distance, a 6-m timed hop test, a triple hop test for distance, a crossover hop test for distance (Noyes et al, 1991). | 6 months postoperatively
Self reported function. | 6 months post operatively
  International Knee Documentation Committee 2000 subjective knee evaluation form.

SECONDARY OUTCOMES:
Pain scores on a visual analog scale | 1 day preoperatively
Degree of swelling measured with The Modified Stroke Test (Logerseth at al, 2010). | 1 day preoperatively
The circumference around the center of the patella will be measured to assess for swelling around the knee joint. | 1 day preoperatively
Passive range of movement compared to the healthy knee, measured with a goniometer. | 1 day preoperatively
Isokinetic muscle strength measured with a fixed dynamometer (isok BI con/con 60/60 240/240 BIODEX) | 1 day preoperatively
Asymmetry in step time between the affected and unaffected leg during down stairs walking. | 1 day preoperatively
  A triaxial kinematic sensor (XSens Mtx) positioned at the level of the lower trunk will be used to identify foot strike and separate left and right steps.
Self reported function | 1 day preoperatively
  International Knee Documentation Committee 2000 subjective knee evaluation form
Muscle atrophy in the quadriceps muscle will be measured 12 and 17 cm above the medial knee joint line. | 1 day preoperatively
Passive range of movement compared to the healthy knee, measured with a goniometer. | at discharge
Pain scores on a visual analog scale. | at discharge
Difficulties with walking downstairs on a visual analog scale. | 1 day preoperative
Pain scores on a visual analog scale. | 6 weeks post operatively
Difficulties with walking down stairs on a visual analog scale. | 6 weeks postoperatively
Degree of swelling measured with The Modified Stroke Test (Logerseth at al, 2010). | 6 weeks postoperatively
The circumference around the center of the patella will be measured to assess for swelling around the knee joint. | 6 weeks postoperatively
Passive range of movement compared to the healthy knee will be measured with a goniometer. | 6 weeks postoperatively
Asymmetry in step time between the affected and unaffected leg during down stairs walking. | 6 weeks postoperatively
  A triaxial kinematic sensor (XSens Mtx) positioned at the level of the lower trunk will be used to identify foot strike and separate left and right steps.
Muscle atrophy in the quadriceps muscle will be measured 12 and 17 cm above the medial knee joint line. | 6 weeks postoperatively
Knee joint laxity measured with knee laxity testing device (KT 1000). | 6 weeks postoperatively
Asymmetry in step time between the affected and unaffected leg during down stairs walking. | 3 months postoperatively
  A triaxial kinematic sensor (XSens Mtx) positioned at the level of the lower trunk will be used to identify foot strike and separate left and right steps.
Pain scores on a visual analog scale. | 3 months postoperatively
Difficulties with walking down stairs on a visual analog scale. | 3 months postoperatively
Degree of swelling measured with The Modified Stroke Test (Logerseth at al, 2010). | 3 months postoperatively
The circumference around the center of the patella will be measured to assess for swelling around the knee joint. | 3 months postoperatively
Passive range of movement compared to the healthy knee, measured with a goniometer. | 3 months postoperatively
Muscle atrophy in the quadriceps muscle will be measured 12 and 17 cm above the medial knee joint line. | 3 months postoperatively
Knee joint laxity measured with a knee laxity testing device (KT 1000). | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Willemijn Vervaat, MSc, Principal Investigator — Haraldsplass Deaconess Hospital
Locations (1):
- Haraldsplass Deaconess hospital, Bergen, Norway

REFERENCES:
- [Background] Adlerton AK, Moritz U, Moe-Nilssen R. Forceplate and accelerometer measures for evaluating the effect of muscle fatigue on postural control during one-legged stance. Physiother Res Int. 2003;8(4):187-99. doi: 10.1002/pri.289. PMID 14730723
- [Background] Arvidsson I, Arvidsson H, Eriksson E, Jansson E. Prevention of quadriceps wasting after immobilization: an evaluation of the effect of electrical stimulation. Orthopedics. 1986 Nov;9(11):1519-28. doi: 10.3928/0147-7447-19861101-08. PMID 3491982
- [Background] Bjordal JM, Arnly F, Hannestad B, Strand T. Epidemiology of anterior cruciate ligament injuries in soccer. Am J Sports Med. 1997 May-Jun;25(3):341-5. doi: 10.1177/036354659702500312. PMID 9167814
- [Background] Daniel DM, Stone ML, Dobson BE, Fithian DC, Rossman DJ, Kaufman KR. Fate of the ACL-injured patient. A prospective outcome study. Am J Sports Med. 1994 Sep-Oct;22(5):632-44. doi: 10.1177/036354659402200511. PMID 7810787
- [Background] de Jong SN, van Caspel DR, van Haeff MJ, Saris DB. Functional assessment and muscle strength before and after reconstruction of chronic anterior cruciate ligament lesions. Arthroscopy. 2007 Jan;23(1):21-8, 28.e1-3. doi: 10.1016/j.arthro.2006.08.024. PMID 17210423
- [Background] Drechsler WI, Cramp MC, Scott OM. Changes in muscle strength and EMG median frequency after anterior cruciate ligament reconstruction. Eur J Appl Physiol. 2006 Dec;98(6):613-23. doi: 10.1007/s00421-006-0311-9. Epub 2006 Oct 12. PMID 17036217
- [Background] Eitzen I, Holm I, Risberg MA. Preoperative quadriceps strength is a significant predictor of knee function two years after anterior cruciate ligament reconstruction. Br J Sports Med. 2009 May;43(5):371-6. doi: 10.1136/bjsm.2008.057059. Epub 2009 Feb 17. PMID 19224907
- [Background] Helbostad JL, Vereijken B, Hesseberg K, Sletvold O. Altered vision destabilizes gait in older persons. Gait Posture. 2009 Aug;30(2):233-8. doi: 10.1016/j.gaitpost.2009.05.004. Epub 2009 May 31. PMID 19487126
- [Background] Hodt-Billington C, Helbostad JL, Moe-Nilssen R. Should trunk movement or footfall parameters quantify gait asymmetry in chronic stroke patients? Gait Posture. 2008 May;27(4):552-8. doi: 10.1016/j.gaitpost.2007.07.015. Epub 2007 Sep 25. PMID 17897830
- [Background] Holder-Powell HM, Di Matteo G, Rutherford OM. Do knee injuries have long-term consequences for isometric and dynamic muscle strength? Eur J Appl Physiol. 2001 Aug;85(3-4):310-6. doi: 10.1007/s004210100474. PMID 11560085
- [Background] Johansson H, Sjolander P, Sojka P. Receptors in the knee joint ligaments and their role in the biomechanics of the joint. Crit Rev Biomed Eng. 1991;18(5):341-68. PMID 2036801
- [Background] Kowalchuk DA, Harner CD, Fu FH, Irrgang JJ. Prediction of patient-reported outcome after single-bundle anterior cruciate ligament reconstruction. Arthroscopy. 2009 May;25(5):457-63. doi: 10.1016/j.arthro.2009.02.014. PMID 19409302
- [Background] McHugh MP, Tyler TF, Browne MG, Gleim GW, Nicholas SJ. Electromyographic predictors of residual quadriceps muscle weakness after anterior cruciate ligament reconstruction. Am J Sports Med. 2002 May-Jun;30(3):334-9. doi: 10.1177/03635465020300030601. PMID 12016072
- [Background] Moe-Nilssen R. A new method for evaluating motor control in gait under real-life environmental conditions. Part 2: Gait analysis. Clin Biomech (Bristol). 1998 Jun;13(4-5):328-335. doi: 10.1016/s0268-0033(98)00090-4. PMID 11415804
- [Background] Moe-Nilssen R. A new method for evaluating motor control in gait under real-life environmental conditions. Part 1: The instrument. Clin Biomech (Bristol). 1998 Jun;13(4-5):320-327. doi: 10.1016/s0268-0033(98)00089-8. PMID 11415803
- [Background] Moe-Nilssen R, Helbostad JL, Akra T, Birdedal L, Nygaard HA. Modulation of gait during visual adaptation to dark. J Mot Behav. 2006 Mar;38(2):118-25. doi: 10.3200/JMBR.38.2.118-125. PMID 16531394
- [Background] Myklebust G, Holm I, Maehlum S, Engebretsen L, Bahr R. Clinical, functional, and radiologic outcome in team handball players 6 to 11 years after anterior cruciate ligament injury: a follow-up study. Am J Sports Med. 2003 Nov-Dec;31(6):981-9. doi: 10.1177/03635465030310063901. PMID 14623667
- [Background] Noyes FR, Barber SD, Mangine RE. Abnormal lower limb symmetry determined by function hop tests after anterior cruciate ligament rupture. Am J Sports Med. 1991 Sep-Oct;19(5):513-8. doi: 10.1177/036354659101900518. PMID 1962720
- [Background] Rice DA, McNair PJ. Quadriceps arthrogenic muscle inhibition: neural mechanisms and treatment perspectives. Semin Arthritis Rheum. 2010 Dec;40(3):250-66. doi: 10.1016/j.semarthrit.2009.10.001. Epub 2009 Dec 2. PMID 19954822
- [Background] Sorsdahl AB, Moe-Nilssen R, Strand LI. Test-retest reliability of spatial and temporal gait parameters in children with cerebral palsy as measured by an electronic walkway. Gait Posture. 2008 Jan;27(1):43-50. doi: 10.1016/j.gaitpost.2007.01.001. Epub 2007 Feb 14. PMID 17300940
- [Background] Young A. Current issues in arthrogenous inhibition. Ann Rheum Dis. 1993 Nov;52(11):829-34. doi: 10.1136/ard.52.11.829. PMID 8250616
- [Background] Heijne A, Ang BO, Werner S. Predictive factors for 12-month outcome after anterior cruciate ligament reconstruction. Scand J Med Sci Sports. 2009 Dec;19(6):842-9. doi: 10.1111/j.1600-0838.2008.00852.x. Epub 2008 Aug 5. PMID 19508651
- [Background] Helbostad JL, Leirfall S, Moe-Nilssen R, Sletvold O. Physical fatigue affects gait characteristics in older persons. J Gerontol A Biol Sci Med Sci. 2007 Sep;62(9):1010-5. doi: 10.1093/gerona/62.9.1010. PMID 17895440
- [Background] Williams GN, Barrance PJ, Snyder-Mackler L, Buchanan TS. Altered quadriceps control in people with anterior cruciate ligament deficiency. Med Sci Sports Exerc. 2004 Jul;36(7):1089-97. doi: 10.1249/01.mss.0000131959.20666.11. PMID 15235310